CLINICAL TRIAL: NCT00088036
Title: Efficacy and Safety of Olanzapine in Patients With Borderline Personality Disorder: A Randomized Double-Blind Comparison With Placebo
Brief Title: Efficacy and Safety of Olanzapine in Patients With Borderline Personality Disorder
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 6253; F1D-MC-HGKK
Record Dates: First submitted 2004-07-19; First posted 2004-07-21 (Estimated); Last update posted 2006-07-24 (Estimated); Status verified 2006-07

CONDITIONS: Borderline Personality Disorder
MeSH Terms: conditions — Borderline Personality Disorder | interventions — Olanzapine

INTERVENTIONS:
Drug: Olanzapine

SUMMARY:
The purpose of the protocol is to evaluate the efficacy and safety of olanzapine compared with placebo in patients with Borderline Personality Disorder (BPD).

ELIGIBILITY:
Inclusion Criteria:

* Patients must be of outpatient status at Visit 1 and through Visit 2
* Patients must be 18 through 65 years of age at Visit 1
* Patients must meet all of the DSM-IV-TR General Diagnostic Criteria for a Personality Disorder AND Patients must meet DSM-IV-TR diagnostic criteria for BPD as determined by the DIPD-IV, confirmed by a psychiatrist with training in the evaluation and assessment of BPD.
* The symptom severity as assessed by the total score of the ZAN-BPD, confirmed by a psychiatrist with training in the evaluation and assessment of BPD, must be greater than or equal to 9 at Visit 2.
* Female patients of childbearing potential must test negative for pregnancy and must be using medically accepted means of contraception throughout the study. Use of any oral or injectable contraception must be initiated prior to Visit 2.

Exclusion Criteria:

* Investigators, study site personnel directly affiliated with the study, or immediate family of investigator site personnel directly affiliated with the study. Immediate family is defined as a spouse, parent, child, or sibling, whether biological or legally adopted.
* Persons employed by Lilly (that is, employees, temporary contract workers, or designees responsible for the conduct of the study). Immediate family of Lilly employees may participate in Lilly-sponsored clinical trials, but are not permitted to participate at a Lilly facility. Immediate family is defined as a spouse, parent, child, or sibling, whether biological or legally adopted
* Have previously participated (have been randomized) or withdrawn from this study or any other Lilly sponsored study investigating olanzapine.
* Have had previous treatment with olanzapine unless, in the opinion of the investigator, the patient's previous treatment was inadequate in dose or duration to provide an accurate assessment of the therapy, or the effect of olanzapine was confounded by concomitant medication.
* Female patients who are either pregnant or nursing.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 450
Dates: Start 2004-02; Study Completion 2006-01

PRIMARY OUTCOMES:
To assess the efficacy of olanzapine therapy (5.0-10.0 mg/day) compared with placebo in patients with BPD,as defined by DSM-IV-TR criteria,
in improving overall symptomatology as measured by the last observation carried forward (LOCF) mean change from baseline to endpoint in the ZAN-BPD total score for up to 12 weeks of double-blind treatment.

SECONDARY OUTCOMES:
To assess the efficacy of olanzapine 2.5 mg/day compared with placebo in patients with BPD, as defined by DSM-IV-TR criteria
in improving overall symptomatology as measured by last observation carried forward (LOCF) mean change from baseline to endpoint in the ZAN-BPD total score for up to 12 weeks of double-blind treatment
to evaluate the level of functioning as measured by LOCF mean change from baseline to endpoint on the Sheehan Disability Scale (Work, Social Life,and Family Life/Home Responsibilities)total score
and individual scores(Work, Social Life,Family Life/Home Responsibilities, Days Lost, and Days Under Productive)
to assess the reduction of aggression, suicidality, and irritability as measured by the LOCF mean change from baseline to endpoint in the rating of the Overt Aggression Scale-Modified (OAS-M) total score
to assess the reduction of self-mutilation determined by the mean frequency of self-mutilation attempts as captured on the Lifetime Self-Destructiveness scale (LSDS), which will measure both frequency and nature of attempts
The frequency of self-mutilation for each patient will be calculated as the number of self-mutilations divided by the patient's total number of study drug exposure
(Self-mutilation is defined as deliberate physical self harm without the intent to commit suicide)
to assess the reduction of suicide attempts as determined by the mean frequency of suicide attempts.
The frequency of suicide attempts for each patient will be calculated as the number of suicide attempts divided by the patient's total number of days of study drug exposure
to assess the treatment of the core domains of BPD as assessed by LOCF mean change from baseline to endpoint in each of the four ZAN-BPD domain scores (cognitive disturbances,disturbed relationships,affective disturbances,and impulsivity)
to assess the following symptom domains (paranoid ideation, psychoticism, anxiety, depression, anger/hostility, interpersonal sensitivity, phobic anxiety, obsessive-compulsive, and somatization)on the Global Severity Index of the SCL-90-R
as determined by the LOCF mean change from baseline to endpoint
to evaluate the rate of response, time in response, and time to response. Levels of response are defined as a 30% and 50% reduction in the ZAN-BPD total score from baseline (Visit 2)
to assess the treatment of depressive mood symptoms as measured by LOCF mean change from baseline to endpoint in the total score on the Montgomery-Asberg Depression Rating Scale (MADRS)
to assess the resource utilization by frequency divided by the patient's total number of days of study drug exposure for days hospitalized for physical and psychological reasons,number of hospital admissions
or medical visits(emergency department, general and special care physicians, and other mental health care professionals
to evaluate the level of functioning in patients as measured by LOCF mean change from baseline to endpoint on the GAF
to assess the safety as measured by treatment-emergency adverse events (TEAE), change in vital signs and laboratory analytes, electrocardiograms and severity of any extrapyramidal symptoms (EPS)
The Simpson Angus Scale, Abnormal Involuntary Movement Scale and Barnes Akathisia Scale will be used to measure EPS
The objectives of Study Period III (Open Label Extension Period are:
to assess the longer term safety of olanzapine for up to 12 additional weeks of therapy
as measured by TEAE, change in vital signs and laboratory analytes, ECG and severity of EPS.
to explore the efficacy of continued olanzapine treatment for up to 12 additional weeks of therapy
as measured by the ZAN-BPD total score, MADRS, Sheehan Disability Scale and LSDS
to assess resource utilization by frequency of divided by the patient's total number of days of study drug exposure for
days hospitalized for physical and psychological reasons, number of hospital admissions
or medical visits (emergency department, general and special care physicians or other mental health care professionals

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (15):
- United States (7):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon-Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, National City, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern time (UTC/GMT - 5 hours, EST), or speak with your personal physician, New Haven, Connecticut
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon-Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, Indianapolis, Indiana
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon-Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, Jackson, Mississippi
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon-Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, The Bronx, New York
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon-Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, Memphis, Tennessee
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon-Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, Houston, Texas
- Argentina (4):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon-Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, Capital Federal, Buenos Aires
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon-Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, La Plata, Buenos Aires
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon-Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, Villa Alberdi, Córdoba Province
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon-Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, Buenos Aires
- Poland (2):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon-Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, Choroszcz
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon-Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, Torun
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon-Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, Bucharest, Sector 4, Romania
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon-Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, Istanbul, Capa, Turkey (Türkiye)

REFERENCES:
- [Derived] Stoffers-Winterling JM, Storebo OJ, Pereira Ribeiro J, Kongerslev MT, Vollm BA, Mattivi JT, Faltinsen E, Todorovac A, Jorgensen MS, Callesen HE, Sales CP, Schaug JP, Simonsen E, Lieb K. Pharmacological interventions for people with borderline personality disorder. Cochrane Database Syst Rev. 2022 Nov 14;11(11):CD012956. doi: 10.1002/14651858.CD012956.pub2. PMID 36375174
- [Derived] Houston JP, Kohler J, Bishop JR, Ellingrod VL, Ostbye KM, Zhao F, Conley RR, Poole Hoffmann V, Fijal BA. Pharmacogenomic associations with weight gain in olanzapine treatment of patients without schizophrenia. J Clin Psychiatry. 2012 Aug;73(8):1077-86. doi: 10.4088/JCP.11m06916. PMID 22967772
- [Derived] Zanarini MC, Schulz SC, Detke HC, Tanaka Y, Zhao F, Lin D, Deberdt W, Kryzhanovskaya L, Corya S. A dose comparison of olanzapine for the treatment of borderline personality disorder: a 12-week randomized, double-blind, placebo-controlled study. J Clin Psychiatry. 2011 Oct;72(10):1353-62. doi: 10.4088/JCP.08m04138yel. PMID 21535995
- [Derived] Houston J, Dharia S, Bishop JR, Ellingrod VL, Fijal B, Jacobson JG, Hoffmann VP. Association of DRD2 and ANKK1 polymorphisms with prolactin increase in olanzapine-treated women. Psychiatry Res. 2011 May 15;187(1-2):74-9. doi: 10.1016/j.psychres.2010.10.020. Epub 2010 Nov 20. PMID 21095016